CLINICAL TRIAL: NCT05855421
Title: Efficacy and Safety of Auricular Acupuncture in Depression During the Covid 19 Pandemic: a Multicenter Triple-blinded Randomized Clinical Trial
Brief Title: Efficacy and Safety of Auricular Acupuncture in Depression During the Covid 19 Pandemic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Sul de Santa Catarina (Other Government)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, DANIEL MAURICIO DE OLIVEIRA RODRIGUES, ND, MSc., Universidade do Sul de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USantaCatarina; 2018/17469-5 (Other Grant/Funding Number: Fundacao de Amparo a Pesquisa do Estado de Sao Paulo)
Record Dates: First submitted 2023-05-10; First posted 2023-05-11 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Depressive Symptoms; Depression; Anxiety; Insomnia; Quality of Life
Keywords: depression; auricular acupuncture; clinical trial; anxiety; insomnia; quality of life
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Acupuncture, Ear; Auriculotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Specific Auricular Acupuncture (Experimental): 12 sessions in 6 weeks, 6 ear points of Chinese Tradicional Medicine - liver, kidney, shenmen, subcortex, heart and lung, with a semi-permanent needle (0,2x2,5mm). Participants will be instructed to stimulate the area 3 times a day.
  Interventions: Device: Auricular Acupuncture
- Inespecific Auricular Acupuncture (Sham Comparator): 12 sessions in 6 weeks, 6 ear points not related to chinese specific points - cheek, outer ear, 4 points non-reactive on the ear helix, with a semi-permanent needle (0,2x1,0mm). Participants will be instructed to stimulate the area 3 times a day.
  Interventions: Device: Auricular Acupuncture

INTERVENTIONS:
Device: Auricular Acupuncture — Aplication of semi-permanents needls in the ear by an experient and specialized professional using tradicional chinese maps and a specific device to find acupuncture points. There is a gap of one day minimum between sessions and two non-consecutive absences are allowed.
  Other Names: Ear Acupuncture; Auriculotherapy

SUMMARY:
Participants with moderate depressive symptoms measured by PHQ-9 will be randomized to receive auricular acupuncture. The triple blinded procedure will be conducted in 12 sessions (6 weeks). The primary outcome is the response to the treatment 3 months after inclusion.

DETAILED DESCRIPTION:
Depression, often under-diagnosed and under-treated, is the leading cause of disability worldwide and contributes significantly to the global burden of diseases, with university students being a major risk group. There is a growing demand for non-pharmacological treatments for depression. In this sense, auricular acupuncture is considered a simple, low cost technique, well accepted by patients. The Unified Health System (Sistema Único de Saúde -SUS) incorporated this practice in 2006, but there is a lack of studies evaluating its efficacy and safety. The main objective of this study is to evaluate the efficacy of auricular acupuncture to reduce depressive symptoms in comparison with usual care and non-specific auricular acupuncture. This is a randomized clinical trial, blinded to the evaluator, participant and statistician. The study sample will be composed of 280 university students, divided equally into two groups: Experimental group - GE (auricular acupuncture) and Control group - GC (non-specific auricular acupuncture). The GE and GC participants will be submitted to 12 sessions of auricular acupuncture, 2 times a week. The primary outcome of the study will be the proportion of participants who present improvement of 50% or more in their symptoms, evaluated by the PHQ-9, three months after inclusion. The secondary outcomes will be: improvement of 50% or more in their symptoms, after six months; quality of life (SF-36), change in the use of antidepressant medication, events and adverse effects, levels of Brain-derived neurotrophic factor (BDNF), Interleukin 1β, Interleukin-6 and TNF-α in blood plasma. The data will be analyzed aiming at treating according to the principles of CONSORT.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years old
* PHQ-9 score between 10 and 19 (moderate depression)
* Availability for sessions

Exclusion Criteria:

Use complementary and integrative practices at the last 3 months; Suicidal risk evaluated by question number 9 in the PHQ-9 Severe depression score in the PHQ-9 Prior use of auricular acupuncture Pregnancy Menopause Tape and metal allergy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male; Female; Non-binary
Enrollment: 280 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Decrease of Depression Symptoms | 3 months
  The efficacy of auricular acupuncture to reduce depression symptoms compared to non-specific auricular acupuncture 3 months after study inclusion.

SECONDARY OUTCOMES:
BDNF, Interleukin, TNF | 6 weeks
  Levels of BDNF, Interleukin 1β, Interleukin-6 and TNF-α, evaluated at the beginning and end of auricular acupuncture applications (end of the sixth week of application)
Decrease of Depression Symptoms | 6 weeks
  The efficacy of auricular acupuncture to reduce depression symptoms compared to non-specific auricular acupuncture 6 weeks after study inclusion.
Decrease of Depression Symptoms | 6 months
  The efficacy of auricular acupuncture to reduce depression symptoms compared to non-specific auricular acupuncture 6 months after study inclusion.
Decrease of Depression Symptoms | 4 weeks
  The efficacy of auricular acupuncture to reduce depression symptoms compared to non-specific auricular acupuncture 4 weeks after study inclusion.
Decrease of Insomnia | 3 months
  The efficacy of auricular acupuncture to reduce insomnia compared to non-specific auricular acupuncture 3 months after study inclusion.
Decrease of Insomnia | 6 months
  The efficacy of auricular acupuncture to reduce insomnia compared to non-specific auricular acupuncture 6 months after study inclusion.
Decrease of Insomnia | 4 weeks
  The efficacy of auricular acupuncture to reduce insomnia compared to non-specific auricular acupuncture 4 weeks after study inclusion.
Decrease of Insomnia | 6 weeks
  The efficacy of auricular acupuncture to reduce insomnia compared to non-specific auricular acupuncture 6 weeks after study inclusion.
Decrease of Anxiety Symptoms | 3 months
  The efficacy of auricular acupuncture to reduce anxiety symptoms compared to non-specific auricular acupuncture 3 months after study inclusion.
Decrease of Anxiety Symptoms | 6 months
  The efficacy of auricular acupuncture to reduce anxiety symptoms compared to non-specific auricular acupuncture 6 months after study inclusion.
Decrease of Anxiety Symptoms | 4 weeks
  The eficacy of auricular acupuncture to reduce anxiety symptoms compared to non-specific auricular acupuncture 4 weeks after study inclusion.
Decrease of Anxiety Symptoms | 6 weeks
  The efficacy of auricular acupuncture to reduce anxiety symptoms compared to non-specific auricular acupuncture 6 weeks after study inclusion.
Increase of Quality of Life | 3 months
  The efficacy of auricular acupuncture to increase quality of life compared to non-specific auricular acupuncture 3 months after study inclusion.
Increase of Quality of Life | 6 months
  The efficacy of auricular acupuncture to increase quality of life compared to non-specific auricular acupuncture 6 months after study inclusion.
Increase of Quality of Life | 4 weeks
  The efficacy of auricular acupuncture to increase quality of life compared to non-specific auricular acupuncture 4 weeks after study inclusion.
Increase of Quality of Life | 6 weeks
  The efficacy of auricular acupuncture to increase quality of life compared to non-specific auricular acupuncture 6 weeks after study inclusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade do Sul de Santa Catarina, Palhoça, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No
There is no IPD to be shared.

REFERENCES:
- [Background] AMERICAN PSYCHIATRIC ASSOCIATION. Diretrizes para o tratamento de transtornos psiquiátricos: compêndio 2006. Porto Alegre: Artmed, 2008.
- [Background] AMERICAN PSYCHIATRIC ASSOCIATION. Manual diagnóstico e estatístico de transtornos mentais: DSM-5. Porto Alegre: Artmed, 2014.
- [Background] BARLOW, D.H; DURAND, V.M. Psicopatologia: uma abordagem integrada. São Paulo: Cengage Learning, 2008.
- [Background] BECK, A.T.; ALFORD, B.A. Depressão causas e tratamento. 2. ed. Porto Alegre: Artmed, 2011.
- [Background] BRASIL. Ministério da Saúde. Secretaria de Atenção à Saúde. Departamento de Atenção Básica. Política Nacional de Práticas Integrativas e Complementares no SUS - PNPIC. Brasília: Ministério da Saúde, 2006.
- [Background] BRASIL. Ministério da Saúde. Secretaria de Atenção à Saúde. Departamento de Atenção Básica. Portaria amplia oferta de PICS. 2019.
- [Background] Brody DJ, Pratt LA, Hughes JP. Prevalence of Depression Among Adults Aged 20 and Over: United States, 2013-2016. NCHS Data Brief. 2018 Feb;(303):1-8. PMID 29638213
- [Background] BROWNER, W.S.; NEWMAN, T.B.; HULLEY, S.G. Estimando o tamanho da amostra e o poder estatístico: aplicações e exemplos. In: HULLER, S.G et al. Delineando a pesquisa clínica: uma abordagem epidemiológica. 3. ed. Porto Alegre: Artmed, 2008.
- [Background] Bus BA, Molendijk ML, Tendolkar I, Penninx BW, Prickaerts J, Elzinga BM, Voshaar RC. Chronic depression is associated with a pronounced decrease in serum brain-derived neurotrophic factor over time. Mol Psychiatry. 2015 May;20(5):602-8. doi: 10.1038/mp.2014.83. Epub 2014 Aug 26. PMID 25155878
- [Background] Cha NH, Park YK, Sok SR. Effects of Auricular Acupressure Therapy on Stress and Sleep Disturbance of Middle-Aged Women in South Korea. Holist Nurs Pract. 2017 Mar/Apr;31(2):102-109. doi: 10.1097/HNP.0000000000000197. PMID 28181975
- [Background] CICONELLI, R.M. et al. Tradução para a língua portuguesa e validação do questionário genérico de avaliação de qualidade de vida SF-36 (Brasil SF-36). Rev Bras Reumatol., v. 29, n. 3, p. 154-50. 1997.
- [Background] COCHRANE COMPLEMENTARY MEDICINE. About us. 2018
- [Background] DAL MAS, Walter Douglas. Acupuntura auricular na doutrina brasileira. São Paulo: Roca, 2004.
- [Background] Ell K, Unutzer J, Aranda M, Gibbs NE, Lee PJ, Xie B. Managing depression in home health care: a randomized clinical trial. Home Health Care Serv Q. 2007;26(3):81-104. doi: 10.1300/J027v26n03_05. PMID 17804354
- [Background] FOCKS, C. Atlas de acupuntura: com sequência de fotos e ilustrações, textos didáticos e indicações clínicas. Barueri: Manole, 2005.
- [Background] Fu WB, Fan L, Zhu XP, He Q, Wang L, Zhuang LX, Liu YS, Tang CZ, Li YW, Meng CR, Zhang HL, Yan J. Depressive neurosis treated by acupuncture for regulating the liver--a report of 176 cases. J Tradit Chin Med. 2009 Jun;29(2):83-6. doi: 10.1016/s0254-6272(09)60037-6. PMID 19663089
- [Background] Geib J, Rieger MA, Joos S, Eschweiler GW, Dresler T, Metzger FG. Introduction of auricular acupuncture in elderly patients suffering from major depression: protocol of a mixed methods feasibility study. Biomed Res Int. 2015;2015:678410. doi: 10.1155/2015/678410. Epub 2015 Apr 15. PMID 25954756
- [Background] Guo N, Robakis T, Miller C, Butwick A. Prevalence of Depression Among Women of Reproductive Age in the United States. Obstet Gynecol. 2018 Apr;131(4):671-679. doi: 10.1097/AOG.0000000000002535. PMID 29528926
- [Background] Hamilton JP, Farmer M, Fogelman P, Gotlib IH. Depressive Rumination, the Default-Mode Network, and the Dark Matter of Clinical Neuroscience. Biol Psychiatry. 2015 Aug 15;78(4):224-30. doi: 10.1016/j.biopsych.2015.02.020. Epub 2015 Feb 24. PMID 25861700
- [Background] Huang W, Pach D, Napadow V, Park K, Long X, Neumann J, Maeda Y, Nierhaus T, Liang F, Witt CM. Characterizing acupuncture stimuli using brain imaging with FMRI--a systematic review and meta-analysis of the literature. PLoS One. 2012;7(4):e32960. doi: 10.1371/journal.pone.0032960. Epub 2012 Apr 9. PMID 22496739
- [Background] Hendrick V, Altshuler L, Cohen L, Stowe Z. Evaluation of mental health and depression during pregnancy: position paper. Psychopharmacol Bull. 1998;34(3):297-9. PMID 9803758
- [Background] King HC, Spence DL, Hickey AH, Sargent P, Elesh R, Connelly CD. Auricular acupuncture for sleep disturbance in veterans with post-traumatic stress disorder: a feasibility study. Mil Med. 2015 May;180(5):582-90. doi: 10.7205/MILMED-D-14-00451. PMID 25939115
- [Background] Ibrahim AK, Kelly SJ, Adams CE, Glazebrook C. A systematic review of studies of depression prevalence in university students. J Psychiatr Res. 2013 Mar;47(3):391-400. doi: 10.1016/j.jpsychires.2012.11.015. Epub 2012 Dec 20. PMID 23260171
- [Background] Irwin MR, Miller AH. Depressive disorders and immunity: 20 years of progress and discovery. Brain Behav Immun. 2007 May;21(4):374-83. doi: 10.1016/j.bbi.2007.01.010. Epub 2007 Mar 13. PMID 17360153
- [Background] Jorm AF, Korten AE, Jacomb PA, Christensen H, Rodgers B, Pollitt P. "Mental health literacy": a survey of the public's ability to recognise mental disorders and their beliefs about the effectiveness of treatment. Med J Aust. 1997 Feb 17;166(4):182-6. doi: 10.5694/j.1326-5377.1997.tb140071.x. PMID 9066546
- [Background] Jorm AF, Medway J, Christensen H, Korten AE, Jacomb PA, Rodgers B. Public beliefs about the helpfulness of interventions for depression: effects on actions taken when experiencing anxiety and depression symptoms. Aust N Z J Psychiatry. 2000 Aug;34(4):619-26. doi: 10.1080/j.1440-1614.2000.00761.x. PMID 10954393
- [Background] Karst M, Winterhalter M, Munte S, Francki B, Hondronikos A, Eckardt A, Hoy L, Buhck H, Bernateck M, Fink M. Auricular acupuncture for dental anxiety: a randomized controlled trial. Anesth Analg. 2007 Feb;104(2):295-300. doi: 10.1213/01.ane.0000242531.12722.fd. PMID 17242083
- [Background] Kessler RC, Soukup J, Davis RB, Foster DF, Wilkey SA, Van Rompay MI, Eisenberg DM. The use of complementary and alternative therapies to treat anxiety and depression in the United States. Am J Psychiatry. 2001 Feb;158(2):289-94. doi: 10.1176/appi.ajp.158.2.289. PMID 11156813
- [Background] Kober A, Scheck T, Schubert B, Strasser H, Gustorff B, Bertalanffy P, Wang SM, Kain ZN, Hoerauf K. Auricular acupressure as a treatment for anxiety in prehospital transport settings. Anesthesiology. 2003 Jun;98(6):1328-32. doi: 10.1097/00000542-200306000-00005. PMID 12766639
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kurebayashi LF, Silva MJ. Efficacy of Chinese auriculotherapy for stress in nursing staff: a randomized clinical trial. Rev Lat Am Enfermagem. 2014 May-Jun;22(3):371-8. doi: 10.1590/0104-1169.3239.2426. PMID 25029046
- [Background] Leung MC, Yip KK, Ho YS, Siu FK, Li WC, Garner B. Mechanisms underlying the effect of acupuncture on cognitive improvement: a systematic review of animal studies. J Neuroimmune Pharmacol. 2014 Sep;9(4):492-507. doi: 10.1007/s11481-014-9550-4. Epub 2014 Jun 6. PMID 24903518
- [Background] Liang Y, Xu B, Zhang XC, Zong L, Chen YL. [Comparative study on effects between electroacupuncture and auricular acupuncture for methamphetamine withdrawal syndrome]. Zhongguo Zhen Jiu. 2014 Mar;34(3):219-24. Chinese. PMID 24843957
- [Background] Liu P, Qin W, Zhang Y, Tian J, Bai L, Zhou G, Liu J, Chen P, Dai J, von Deneen KM, Liu Y. Combining spatial and temporal information to explore function-guide action of acupuncture using fMRI. J Magn Reson Imaging. 2009 Jul;30(1):41-6. doi: 10.1002/jmri.21805. PMID 19557845
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] LUZ, M.T. Cultura Contemporânea e Medicinas Alternativas: Novos paradigmas em saúde no fim do século XX. Physis: Revista Saúde Coletiva. Rio de Janeiro, 15(Suplemento):145-176, 2005.
- [Background] MacPherson H, Thomas K, Walters S, Fitter M. The York acupuncture safety study: prospective survey of 34 000 treatments by traditional acupuncturists. BMJ. 2001 Sep 1;323(7311):486-7. doi: 10.1136/bmj.323.7311.486. No abstract available. PMID 11532841
- [Background] Molendijk ML, Spinhoven P, Polak M, Bus BA, Penninx BW, Elzinga BM. Serum BDNF concentrations as peripheral manifestations of depression: evidence from a systematic review and meta-analyses on 179 associations (N=9484). Mol Psychiatry. 2014 Jul;19(7):791-800. doi: 10.1038/mp.2013.105. Epub 2013 Aug 20. PMID 23958957
- [Background] NATIONAL INSTITUTE OF MENTAL HEALTH. Depression and College Students. 2018. https://www.nimh.nih.gov/health/publications/depression-and-collegestudents/index.shtml
- [Background] PRADO, J.M. Aplicação da acupuntura auricular verdadeira e sham no tratamento do estresse em enfermeiros. 2014. 98 p. Dissertação (Mestrado em Enfermagem na Saúde do adulto), Universidade de São Paulo, São Paulo, 2014.
- [Background] Raison CL, Capuron L, Miller AH. Cytokines sing the blues: inflammation and the pathogenesis of depression. Trends Immunol. 2006 Jan;27(1):24-31. doi: 10.1016/j.it.2005.11.006. Epub 2005 Nov 28. PMID 16316783
- [Background] SABBAG, S.H.F. et al. A. Origem e desenvolvimento da Naturologia no Brasil: aspectos conceituais, históricos e políticos. Cad. Naturol. Terap. Complem, v. 6, n. 11, p. 59-68, Set. /Abr., 2017.
- [Background] Santos IS, Tavares BF, Munhoz TN, Almeida LS, Silva NT, Tams BD, Patella AM, Matijasevich A. [Sensitivity and specificity of the Patient Health Questionnaire-9 (PHQ-9) among adults from the general population]. Cad Saude Publica. 2013 Aug;29(8):1533-43. doi: 10.1590/0102-311x00144612. Portuguese. PMID 24005919
- [Background] Set T, Cayir Y, Pirim AB. Effects of ear acupuncture therapy for obesity on the depression of obese women. Acupunct Med. 2014 Oct;32(5):427-9. doi: 10.1136/acupmed-2014-010626. Epub 2014 Aug 6. PMID 25098839
- [Background] Simon NM, McNamara K, Chow CW, Maser RS, Papakostas GI, Pollack MH, Nierenberg AA, Fava M, Wong KK. A detailed examination of cytokine abnormalities in Major Depressive Disorder. Eur Neuropsychopharmacol. 2008 Mar;18(3):230-3. doi: 10.1016/j.euroneuro.2007.06.004. Epub 2007 Aug 3. PMID 17681762
- [Background] Smith CA, Armour M, Lee MS, Wang LQ, Hay PJ. Acupuncture for depression. Cochrane Database Syst Rev. 2018 Mar 4;3(3):CD004046. doi: 10.1002/14651858.CD004046.pub4. PMID 29502347
- [Background] SOUZA, F.G.M. Tratamento da depressão. Rev. Bras. Psiquiatr, v. 21, n.1, Maio.1999.
- [Background] STUX, G. BIRCH, S. Padrões de tratamento por acupuntura propostos para estudos clínicos. In: STUX, G. BERMAN, B; POMERANZ, B. Basics of acupuncture. Berlin: Springer, 2005.
- [Background] White A, Hayhoe S, Hart A, Ernst E; BMAS and AACP. British Medical Acupuncture Society and Acupuncture Association of Chartered Physiotherapists. Survey of adverse events following acupuncture (SAFA): a prospective study of 32,000 consultations. Acupunct Med. 2001 Dec;19(2):84-92. doi: 10.1136/aim.19.2.84. PMID 11829164
- [Background] WORLD HEALTH ORGANIZATION. Benchmarks for training in traditional /complementary and alternative medicine: benchmarks for training in traditional Chinese medicine. 2010. Genebra: Who: 2010.
- [Background] WORLD HEALTH ORGANIZATION. WHO Traditional Medicine Strategy 2014-2023. Genebra: WHO. 2013.
- [Background] WORLD HEALTH ORGANIZATION. Atlas de Medicina Complementares e Tradicional. 2014. Genebra: OMS.
- [Background] WORLD HEALTH ORGANIZATION. Depression and Other Common Mental Disorders: Global Health Estimates. Genebra: OMS, 2017a.
- [Background] WORLD HEALTH ORGANIZATION. Mental Health. Depression: let's talk. 2017b
- [Background] Lv X, Wang B, Chen Jianbin, Ye J. [Clinical observation of depression after breast cancer operation treated with aurieular point sticking therapy]. Zhongguo Zhen Jiu. 2015 May;35(5):447-50. Chinese. PMID 26255515
- [Background] Zhong LL, Kun W, Lam TF, Zhang SP, Yang JJ, Ziea TC, Ng B, Bian ZX. The combination effects of body acupuncture and auricular acupressure compared to sham acupuncture for body weight control: study protocol for a randomized controlled trial. Trials. 2016 Jul 25;17(1):346. doi: 10.1186/s13063-016-1458-2. PMID 27457720
- [Derived] de Oliveira Rodrigues DM, Menezes PR, Machado Ribeiro Silotto AE, Heps A, Pereira Sanches NM, Schveitzer MC, Faisal-Cury A. Efficacy and Safety of Auricular Acupuncture for Depression: A Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2345138. doi: 10.1001/jamanetworkopen.2023.45138. PMID 38032640

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT05855421/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT05855421/ICF_001.pdf